CLINICAL TRIAL: NCT02485015
Title: The Randomized, Controlled, Multicenter Clinical Trial of Apatinib Plus CIK as the Third Line Therapy for Patients With Advanced Gastric Cancer
Brief Title: The Study of Apatinib Plus CIK as the Third Line Therapy for Patients With Advanced Gastric Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First People's Hospital of Changzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CZYY-GAS-001
Record Dates: First submitted 2015-06-24; First posted 2015-06-30 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Stomach Neoplasms
Keywords: CIK; gastric cancer; Apatinib
MeSH Terms: conditions — Stomach Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apatinib alone (Other): Apatinib(YN968D1) ,850mg,p.o.,qd,continuous.Patients undergo Apatinib.
  Interventions: Drug: Apatinib
- Apatinib+CIK (Experimental): Apatinib(YN968D1) ,850mg,p.o.,qd,continuous. plus autologous cytokine-induced killer cells 3 cycles,every 1 year,continuous.
  Interventions: Biological: Cytokine-Induced Killer Cells; Drug: Apatinib

INTERVENTIONS:
Biological: Cytokine-Induced Killer Cells — Cytokine-Induced Killer Cells are used to treat advanced gastric cancer patients with Apatinib.
  Other Names: CIK
  Arms: Apatinib+CIK
Drug: Apatinib — Advanced gastric cancer patients take Apatinib 850mg qd by mouth.
  Other Names: YN968D1

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Apatinib combined with cytokine-induced killer cell (CIK) vs Apatinib as the third line therapy for patients with advanced gastric cancer.

DETAILED DESCRIPTION:
400 patients with stage Ⅳ Gastric Cancer,who had received surgery and chemotherapy,will be randomly divided into group A（receive Apatinib and CIK treatment ) or group B（just receive Apatinib),and the randomize ratio will be 1:1. Patients in group A will receive 3 cycles of CIK treatment (every 1 year) and Apatinib (continuous).Patients in group B will receive only Apatinib (continuous) .

ELIGIBILITY:
Inclusion Criteria:

* Patients who can accept curative operations 18-70 years old
* Histologically confirmed with gastric cancer at stage Ⅳ
* Patients who can accept oral drugs;
* Eastern Cooperative Oncology Group (ECOG) performance status was 0 - 1.

Exclusion Criteria:

* Hemoglobin<8.0 g/dL,White blood cell <3 X 10^9/L;Platelet count <75 X 10^9/L; alanine aminotransferase, glutamic-oxalacetic transaminase, blood urine nitrogen and creatinine more than normal limits on 3.0 times
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Pregnant or lactating patients
* Known history of Human Immunodeficiency Virus (HIV), Hepatitis C Virus (HCV) or TreponemaPallidun (TP) infection
* Patients who are suffering from serious autoimmune disease
* Patients who had used long time or are using immunosuppressant
* Patients who had active infection
* Patients who are suffering from serious organ dysfunction
* Patients who are suffering from other cancer
* Other situations that the researchers considered unsuitable for this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06; Primary Completion 2030-06 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival(OS) | 3 months

SECONDARY OUTCOMES:
Disease-free survival | 3 months

OTHER OUTCOMES:
Adverse events | 1 months